CLINICAL TRIAL: NCT03650075
Title: A Phase I Study to Determine Safety and Tolerability of MG-S-2525 and to Evaluate Its Pharmacokinetic Profile in Healthy Volunteers
Brief Title: To Determine Safety and Tolerability of MG-S-2525 and to Evaluate Its PK Profile in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Metagone Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MEOMGSA20180103
Record Dates: First submitted 2018-08-20; First posted 2018-08-28 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (SAD) (Placebo Comparator)
  Interventions: Drug: MG-S-2525
- Multiple Ascending Dose (MAD) (Placebo Comparator)
  Interventions: Drug: MG-S-2525
- Food Effect Part (Experimental)
  Interventions: Drug: MG-S-2525

INTERVENTIONS:
Drug: MG-S-2525 — The investigational product is MG-S-2525, which is an oral, small-molecule, anti-inflammatory agent. MG-S-2525 is being developed by Metagone Biotech Inc. and contains the new molecular entity HL0, an inhibitor of MAP3K19 which is up-regulated in disease pathobiology and in response to inflammatory stimuli in IPF.

SUMMARY:
This is a Phase I stage to investigate the safety and tolerability of MG-S-2525 in healthy volunteers. The proposed trial consists of 3 study parts to be conducted at Tri-Service General Hospital and includes Single Ascending Dose (SAD), Multiple Ascending Dose (MAD) and Food Effect parts. This study will enroll up to 16 evaluable subjects in the SAD part, 36 evaluable subjects in the MAD part and enroll up to 20 evaluable subjects for the Food Effect part.

ELIGIBILITY:
Inclusion Criteria:

Single ascending dose (SAD), Multiple ascending dose (MAD) and Food Effect Parts:

1. Healthy male volunteers
2. Subject's age is no less than 20 years old
3. Subjects whose body mass index (BMI) at screening is within a range of ≥18.5 kg/m2 and <25.0 kg/m2.

   BMI = Body Weight (kg) / [Height (m)]2 Body weight is not less than 50 kg
4. Subjects who are judged to be in good health by the investigator based upon the results of physical examinations, chest X-ray (within 180 days prior to the first dose of the study) and routine laboratory tests.
5. Subjects did not take any of the following medications in the specified durations:

   * Any systemically-absorbed medication (excluding vitamins, food supplements, and hormone contraceptives for birth control) within 14 days prior to the first dose of the study
   * Any enzyme inducer/inhibitor and/or known hepatic or renal clearance-altering agents (e.g., erythromycin, cimetidine, barbiturates, phenothiazine, clarithromycin, troleandomycin, ketoconazole, miconazolem fluconazole, itraconazole) within 30 days prior to the first dose of the study
6. Subjects are willing to comply with protocol-stated requirements, instructions and restrictions, followed by understanding and signing the written informed consent form.

   Extra Criteria for the MAD and Food Effect Parts
7. Healthy female volunteers whose body weight is not less than 45 kg
8. Female subjects show negative pregnancy test results within 30 days prior to the first study dose.
9. Female subjects of child-bearing potential, committing to practicing sexual abstinence or using and continue to use a medically acceptable form of birth control for at least 1 month prior to screening (that period will extend to 3 months for oral contraceptive use) and for at least 30 days after the last dose of study drug. For a subject to be considered not to be of child-bearing potential, she must have been amenorrheic for at least 2 years, or must have had a hysterectomy, a bilateral tubal ligation, and/or a bilateral oophorectomy (as determined by the medical history). The male partner of a female study subject with childbearing potential must use a condom and ensure that his partner uses a suitable method of contraception as outlined above.

   Extra Criteria for the MAD Part
10. Subjects who are self-reporting current smokers (>10 pack/years).

Exclusion Criteria:

SAD, MAD and Food Effect Parts:

1. Subjects with any properly diagnosed disease within 30 days prior to the first dose of the study.
2. Subjects with a clinically significant hematological, endocrine, cardiovascular, hepatic, renal, gastrointestinal, and/or pulmonary disorder; subjects with any predisposing condition that might interfere with the absorption, distribution, metabolism and excretion of drugs; subjects who has had any previous gastrointestinal surgery, except appendectomy if performed >90 days prior to the first dose of the study
3. Subjects had participated in investigational drug trials and took any investigational drug within 60 days prior to the first dose of the study.
4. Subjects had blood donation of more than 250 and 500 mL within 60 and 90 days, respectively prior to the first dose of the study.
5. Subjects had a history of drug abuse or alcohol abuse according to the Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria.
6. Subject's medical history shows contraindications or hypersensitivity to the use of test medications [HL0 or any component of drug products].
7. Subjects who have been tested positive for the following tests:

   * Human immunodeficiency virus (HIV)
   * Hepatitis B virus (HBV)
   * Hepatitis C virus (HCV)
8. Subjects who cannot stop caffeine-intake for 48 hours prior to the first study dose and during the entire study period.
9. Subjects with underlying medical, mental or psychological conditions that would impair treatment compliance, or in the opinion of the investigator would not permit to participate in the study
10. Subjects who have received or are taking any medications that may interfere the assessment [e.g., anti-inflammatories, anti-asthma/COPD (chronic obstructive pulmonary disease) and anti-IPF (idiopathic pulmonary fibrosis) medications] for a period of up to 14 days prior to the first dose of the study Extra Criteria for the MAD and Food Effect Parts
11. Female subjects who are lactating Extra criteria for the MAD part
12. Subjects who did not smoke for more than 2 days prior to the first dose of the study or during the study period

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose (MTD) (Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) parts) | approximately 3 weeks (SAD part) or 15 days (MAD part)
  MTD will be determined by study definition
dose limiting toxicity (DLT) (Single Ascending Dose (SAD) and Multiple Ascending Dose (MAD) parts) | approximately 3 weeks (SAD part) or 15 days (MAD part)
  Number of subjects with DLT will be presented by dose group.
total exposure by area under the curve (AUC) (Food Effect Part) | 10 days
  The 90% confidence intervals for geometric mean ratios of Cmax will be estimated and presented by gender.
peak concentration (Cmax) under fasting/fed condition (Food Effect Part) | 10 days
  The 90% confidence intervals for geometric mean ratios of AUC0→inf will be estimated and presented by gender.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No